CLINICAL TRIAL: NCT07317869
Title: Impact Evaluation of the Therapeutic Initiative's Prescribing Portrait and Therapeutics Letter on Opioid Use by Dentists for Dental Pain
Brief Title: Impact Evaluation of the Therapeutic Initiative's Prescribing Portrait and Therapeutics Letter on Opioid Use by Dentists
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government)
Responsible Party: Principal Investigator, Colin Dormuth, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: H25-03753
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Clinical Audit; Quality Improvement; Opioid; Dentistry
Keywords: Randomized controlled trial; Prescribing feedback; Quality improvement; Opioid

STUDY DESIGN:
Intervention Model Description: Investigators randomized actively practicing dentists into three groups, n = 1166 in each group. Groups 1 will receive the "regular" intervention and Group 2 will receive the "enhanced" intervention materials on January 6 2026, while Group 3 will serve as a delayed control and will receive the "regular" intervention 12 months after Groups 1 and 2.
Who Masked: Participant
Masking Description: Dentists will not be masked to their group allocation but will not be aware of the trial arm variations being evaluated or the analytical approach. The statistical analysis plan is being developed by an evaluation committee who are masked to the trial arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Group 1) - Regular intervention bundle (Experimental): Arm A/Group 1 receives the "regular" intervention bundle.
  Interventions: Behavioral: Regular intervention
- Arm B (Group 2) - Enhanced intervention (Experimental): Arm B/Group 2 receives the "enhanced" intervention bundle
  Interventions: Behavioral: Enhanced intervention
- Arm C (Group 3) - Delayed control (Experimental): Arm C/Group 3 is a delayed control group that receives the "regular" intervention materials 12 months after the Arm A and B receive their interventions.
  Interventions: Behavioral: Regular intervention

INTERVENTIONS:
Behavioral: Regular intervention — The "regular" intervention bundle consists of a personalized prescribing "Portrait" showing dentists their opioid prescribing volume and duration over the past five years compared with the provincial median. The Portrait is accompanied by a Therapeutics Letter summarizing evidence-based recommendations for dental pain management, emphasizing that NSAIDs with or without acetaminophen provide similar or better pain control than opioids and are associated with fewer adverse events. Dentists also receive a patient education handout addressing common questions about opioid use for dental pain.
  Arms: Arm A (Group 1) - Regular intervention bundle; Arm C (Group 3) - Delayed control
Behavioral: Enhanced intervention — For the "enhanced" intervention bundle, dentists receive all components of the regular intervention, plus and invitation to participate in facilitated peer audit-and-feedback group sessions to review prescribing data, identify practice gaps, develop improvement strategies, and commit to change. Participants also receive an updated personalized Portrait (updated data) at approximately six months, followed by additional facilitated sessions to review new data and reassess practice enhancement strategies.
  Arms: Arm B (Group 2) - Enhanced intervention

SUMMARY:
The aim of this study is to estimate the impact of providing personalized prescribing data and educational materials on opioid prescribing to dentists in British Columbia, Canada.

The main research questions are:

1. What is the impact of an intervention on the use of opioids for dental pain? The intervention includes a personalized prescribing report (a "Portrait"), brief educational summary, and patient education materials; and
2. Does the impact of the intervention increase when dentists are also invited to attend facilitated audit-and-feedback group sessions and to develop a practice improvement plan? Using administrative health data, the prescribing of those in different combinations of materials in the Early Group will be compared to those in the Delayed Group to estimate the impact of the materials on prescribing by the dentists.

DETAILED DESCRIPTION:
Audit and feedback is a well-established strategy for improving the quality of care in primary healthcare settings. It involves the systematic collection and analysis of healthcare data, followed by the provision of information to healthcare providers to improve the quality of care.

Medical overprescribing of opioids significantly contributed to overdose deaths from 1995-2015. Although illicit synthetic opioids now dominate the overdose crisis, prescription opioids remain implicated in 22% of overdoses and 2% of fatal overdoses in British Columbia (BC). Dentists play an important role in opioid exposure: opioids may be prescribed in up to half of dental procedures, and general dentists account for 13% of all opioid prescriptions in BC.

Based in British Columbia, Canada, the Therapeutics Initiative's Portrait program provides clinicians with individualized prescribing data compared with their peers, paired with evidence-based messaging, and a concise statement summarizing the desired change in prescribing behavior. The Portrait program implements a series of pragmatic trials to improve prescribing where clinicians are randomized into an early intervention and a delayed control group.

This study examines the impact of prescribing Portraits on opioid prescribing by dentists in British Columbia. The Portrait title is "Do you manage dental pain with opioids?" and is accompanied by a Therapeutics Letter entitled "Pharmacological management of dental pain and inflammation."

3,498 active dentists in BC will be randomized into 3 Groups/Arms (n=1166 in each Group) for this intention-to-treat analysis.

On Jan 6, 2026 dentists in Groups 1 and 2 will be mailed their intervention bundles (Group 1 the regular intervention and Group 2 the enhanced intervention). Six months later clinicians in Group 2 will receive a repeat of the enhanced intervention, and 6 months after that (12 months after the first intervention), Group 3 (delayed control group) will receive the regular intervention bundle. The analysis will assess whether the materials led dentists in Groups 1 and 2 to change how they prescribe.

Analysis will be conducted using secondary data from administrative databases from the BC Ministry of Health (under an Information Sharing Agreement). The data are patient level and include anonymized information about demographics, health costs, physician billing codes, prescriptions, outpatient records, and hospitalizations. The data do not include personally identifiable patient information.

The trial will include two primary comparisons: (1) dentists randomized to either intervention arm (regular or enhanced intervention) versus dentists randomized to the control arm, and (2) dentists randomized to the regular intervention versus the enhanced intervention. All analyses will be conducted according to the intention-to-treat principle, with participants analyzed in the groups to which they were originally randomized, regardless of intervention exposure or adherence. In addition to primary outcome measures, the analyses will identify baseline characteristics of dentists and patients by study group (age, age groups, sex, urban vs rural) and monthly opioid prescribing trends for all BC dentists from 12 months prior to release of the materials. This will illustrate background trends in prescribing patterns.

Prescribing outcomes will be analyzed using generalized linear mixed models with a negative binomial distribution to account for overdispersion in count data. Models will estimate rate differences and rate ratios between trial arms over time. Random effects will be included to account for repeated observations within included dentists, and 95% confidence intervals will be adjusted for clustering of patients within included dentists. Time will be modeled explicitly to assess changes in prescribing rates before and after intervention implementation.

Prespecified subgroup analyses will include incident opioid prescribing among opioid-naïve patients. Opioid naïve will be defined using a one-year look-back period with no opioid prescriptions prior to the index dental visit (January 5, 2025 to January 5, 2026).

In addition, based on prior evidence from a large Veterans Affairs study demonstrating an association between high antibiotic prescribing and high opioid prescribing among dentists (adjusted odds ratio 8.40, 95% CI 6.00-11.76), the investigators will conduct a prespecified subgroup analysis examining the association between changes in opioid prescribing and changes in antibiotic prescribing following the research team's prior antibiotic prescribing intervention.

ELIGIBILITY:
Inclusion Criteria:

Dentists will be eligible to receive an individual prescribing Portrait if they meet all of the following criteria:

* Registered with the British Columbia Medical Services Plan (MSP) as being in active practice;
* Have a valid mailing address in British Columbia; and
* Issued ≥10 prescriptions dispensed at community pharmacies between January 5, 2025 and January 5, 2026, as identified in PharmaNet claims data.

Patients will be eligible for inclusion if they meet all of the following criteria:

* Received an opioid prescription from an eligible dentist during the study period (January 6, 2026 to January 6, 2027);
* The opioid prescription was issued by a dentist; and
* Were continuously enrolled in the British Columbia Medical Services Plan (MSP) during the 12 months prior to the opioid prescription.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

* Had a medication dispensed under Plan P in the 12 months prior to the opioid prescription; or
* Filled a prescription for opioid agonist therapy (OAT) within 180 days prior to the opioid prescription.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3498 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2027-01-06 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The number of opioid prescriptions per dentist | From baseline to 12 months post interventions. The baseline is the 12-month period before the date when the prescriber is mailed the intervention bundle.
  The primary outcome is the change from baseline in the number of opioid prescriptions per dentist. The primary measures of effect will be absolute differences between trial arms, differences in prescribing trends over time, and difference-in-differences estimates comparing the intervention period with the pre-intervention period.
Total morphine milligram equivalents (MME) prescribed per dentist | From baseline to 12 months post interventions. The baseline is the 12-month period before the date when the prescriber is mailed the intervention bundle.
  The primary outcome is the change from baseline in the total morphine milligram equivalents (MME) prescribed per dentist. The primary measures of effect will be absolute differences between trial arms, differences in prescribing trends over time, and difference-in-differences estimates comparing the intervention period with the pre-intervention period.

SECONDARY OUTCOMES:
Rate ratios between trial arms | From baseline to 12 months post intervention. The baseline is the 12-month period before the date when the prescriber is mailed the intervention bundle.
  Secondary measures of effect will include relative measures (rate ratios) comparing trial arms.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, ScD, Principal Investigator — University of British Columbia
Locations (1):
- Therapeutics Initiative - Dept of Anesthesiology, Pharmacology & Therapeutics, Faculty of Medicine, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Our data access agreement does not permit sharing of IPD